CLINICAL TRIAL: NCT01352923
Title: Study of Polymorphisms in pear1 Gene Link to Platelet Activation and Signaling Pathway Variations
Status: Withdrawn | Type: Observational
Why Stopped: no resources
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: B322201111373
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2011-05

CONDITIONS: Platelet Function
Keywords: PEAR1 gene; PEAR 1 gene
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- peripheral blood: healthy voluntary donors
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test — preparation of blood platelets

SUMMARY:
In this study PEAR1 polymorphisms effects will be analyze in blood platelets to determine how PEAR1 regulates platelet activation.

DETAILED DESCRIPTION:
Several large-scale studies have confirmed the long held notion that platelet responses to different agonists are highly variable, within well defined populations of healthy donors. Single nucleotide polymorphisms in genes encoding platelet proteins can explain the wide range of responses to standard platelet agonists. Yet, numerous SNPs point towards proteins with previously unknown function in platelets, wich modulate the complex network of signaling events that regulate platelet function and further augment variability. PEAR1 is mainly expressed in platelets and endothelial cells. A few studies have linked SNPs in PEAR1 with decreased or increased platelet responses to various agonists. However, hitherto, no direct functional studies have been carried out to determine whether and how PEAR1 modulate intracellular signaling pathways relevant for platelet function.

ELIGIBILITY:
Inclusion Criteria:

* healthy voluntary donors

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy voluntary donors
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Hoylaerts, Principal Investigator — KU Leuven
Locations (1):
- KUleuven/UZ Gasthuisberg, Leuven, Vlaams Brabant, Belgium